CLINICAL TRIAL: NCT07096037
Title: Evaluation of Safety and Efficacy of Urtica Dioica Cataplasm in the Management of Osgood-Schlatter Disease in Young Athletes: A Study Protocol for Randomized, Double-blind, Placebo Controlled Clinical Trial
Brief Title: Safety and Efficacy of Urtica Dioica Cataplasm in the Management of Osgood-Schlatter Disease in Young Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Amira Zairi, Professor, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDC-OSD-2025
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Osgood-Schlatter Disease
Keywords: Urtica dioica; Osgood-Schlatter disease; KOOS-Child; Visual Analogue Scale
MeSH Terms: conditions — Osteochondrosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Urtica dioica cataplasm (Experimental): Topical application of Urtica dioica cataplasm
  Interventions: Other: Urtica dioica cataplasm
- Standard Care Group (Active Comparator): Oral vitamin D supplementation and physical rest
  Interventions: Drug: Vitamin D; Behavioral: Resting conditions
- Placebo (Placebo Comparator): Topical application of a placebo cataplasm
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Urtica dioica cataplasm — Participants will receive a warm Urtica dioica cataplasm applied topically on the affected knee, once daily for 60 minutes, three times per week (on alternate days) over a 6-week period.
  Arms: Urtica dioica cataplasm
Other: Placebo — Participants will receive a placebo cataplasm, matched in texture, color, and odor to the active treatment. The placebo is inert and safe for pediatric topical use.
  Arms: Placebo
Drug: Vitamin D — Participants will receive oral vitamin D.
  Arms: Standard Care Group
Behavioral: Resting conditions — Reduction in physical activity based on orthopedic advice.
  Arms: Standard Care Group

SUMMARY:
The primary objective of this clinical trial is to evaluate the efficacy and safety of a topical Urtica dioica cataplasm in managing knee pain and functional limitations in athletic children diagnosed with Osgood-Schlatter Disease. Efficacy will be assessed through changes in knee pain using the Visual Analog Scale (VAS) and functional outcomes using the Knee Injury and Osteoarthritis Outcome Score (KOOS). Three groups will be tested:

* UDC Group: topical application of Urtica dioica cataplasm
* Standard Care Group: oral vitamin D supplementation and physical rest
* Placebo Group: topical application of a placebo cataplasm using Beta vulgaris subsp. cicla

ELIGIBILITY:
Inclusion Criteria:

* Healthy male children between 7 and 15 years of age
* Active in regular sports practice (e.g., football)
* Clinically confirmed diagnosis of OSD

Exclusion Criteria:

* Known allergy to Urtica dioica
* Presence of dermatological conditions or lesions on the knees
* Recent use of anti-inflammatory medications
* History of immune or chronic inflammatory diseases
* Diagnosis of any other bone disorder

Ages: 7 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At each clinical visit during the intervention period (three times a week during 6 weeks).
  measured using the Visual Analog Scale (VAS), a 10-cm line anchored by "no pain" (0) and "worst imaginable pain" (10). VAS scores will be recorded at each clinical visit during the intervention period.

SECONDARY OUTCOMES:
Functional knee status | Assessments will be done at baseline and after 6 weeks.
  assessed using the KOOS-Child questionnaire, covering five subscales (pain, symptoms, activities of daily living, sport/recreation function, and knee-related quality of life). Scores range from 0 (extreme dysfunction) to 100 (no symptoms).
Return to sport | 6 weeks
  defined as the number of days post-treatment needed to resume regular athletic activity.

OTHER OUTCOMES:
Adverse events | At each follow-up visit during 6 weeks
  Adverse events (skin reactions, discomfort, or other clinical complaints) will be recorded systematically.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Zairi, Study Director — Department of Biochemistry, Faculty of Medicine of Sousse, University of Sousse, Tunisia; Sahbi El Mtaoua, Principal Investigator — Department of Physical Medicine and Rehabilitation, Hospital Ibn Jazzar of Kairouan, University of Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No